CLINICAL TRIAL: NCT01646203
Title: Phase 1 Study of Anti-TGFβRII Monoclonal Antibody IMC-TR1 (LY3022859) in Patients With Advanced Solid Tumors That Have Failed Standard Therapy or for Which No Standard is Available
Brief Title: A Study of IMC-TR1 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14549; I5I-IE-JTCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-11; First posted 2012-07-20 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms; Tumor
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — LY3022859

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-TR1 (Experimental): Part A - Dose Escalation:
  Cohort 1A: 1.25 mg/kg, intravenously (IV), every 2 weeks of the 6-week treatment cycle
  Cohorts 1B-9: Dose Escalation from 12.5 mg to 1600 mg (flat dose), intravenously (IV), every 2 weeks of the 6-week treatment cycles
  Cohorts 10-12: Dose escalation from 800 mg to 1600 mg (flat dose), intravenously (IV), weekly during the 6-week treatment cycles
  Part B - Disease Specific Cohort Expansion:
  Participants will be enrolled into each of three tumor-specific cohort expansions. Participants will be treated with recommended Phase 2 dose.
  Interventions: Biological: IMC-TR1

INTERVENTIONS:
Biological: IMC-TR1 — Administered intravenously
  Other Names: LY3022859

SUMMARY:
A study to evaluate the safety and tolerability of anti-TGFβRII monoclonal antibody (IMC-TR1) in participants with advanced solid tumors, as well as gather evidence of anti-tumor activity.

DETAILED DESCRIPTION:
This is the first-in-human Phase 1 study of IMC-TR1.

ELIGIBILITY:
Inclusion Criteria:

* Part A and Part B: Participants must be appropriate candidates for experimental therapy, with a solid tumor that has failed standard therapy or for which no standard therapy is available, and evidence of progressive disease

  * Part A only: Participants must have histological or cytological evidence of a solid tumor which is advanced and/or metastatic
  * Part B only: Participants who have failed first-line therapy/standard of care and have histological or cytological evidence of a cancer type for which evidence of activity was observed during Part A or for which preclinical evidence of potential activity has been observed
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1)

  * Part A only: Participants may have measurable or nonmeasurable disease
  * Part B: Participants must have measurable disease
* Have adequate organ function including: Hematologic, Hepatic, Albumin, Coagulation and Renal function
* Have a performance status of ≤ 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued previous treatments for cancer and recovered from the acute effects of therapy
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug
* Females with child bearing potential must have had a negative serum pregnancy test and must not be breastfeeding
* Have an estimated life expectancy that is > 3 months

Exclusion Criteria:

* Have clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months prior to study entry, unstable angina pectoris, congestive heart failure, or uncontrolled hypertension
  * Major electrocardiogram (ECG) abnormalities
  * Major abnormalities documented by echocardiography with Doppler
  * Have known predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress
  * Have Corrected QT Interval (QTc interval) of > 500 msec on screening ECG
* Have other known serious pre-existing medical conditions
* Have received prior investigational therapy targeting Transforming growth factor beta (TGFβ) or its receptors
* Have a known sensitivity to monoclonal antibodies or other therapeutic proteins, to agents of similar biologic composition as IMC-TR1
* Have a high risk of gastrointestinal bleeding, active inflammatory bowel disease, or chronic steroid use
* Are currently using or has received a systemic thrombolytic agent within 28 days prior to enrollment
* Are receiving:

  * full-dose warfarin
  * intravenous heparin or low-molecular-weight heparin
  * chronic daily treatment with aspirin at a dose greater than 325 mg per day or nonsteroidal anti-inflammatory medications known to inhibit platelet function
* Have evidence of retinal disease or are a monocular participant
* Have received a solid organ transplant, bone marrow transplant or stem cell transplant
* Have symptomatic central nervous system (CNS) malignancy or untreated metastasis
* Have acute or chronic leukemia
* Have a known active fungal, bacterial, and/or viral infection including human immunodeficiency virus or viral hepatitis requiring treatment
* Has a positive fecal occult blood test within 14 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Antonio, Texas

REFERENCES:
- [Derived] Tolcher AW, Berlin JD, Cosaert J, Kauh J, Chan E, Piha-Paul SA, Amaya A, Tang S, Driscoll K, Kimbung R, Kambhampati SR, Gueorguieva I, Hong DS. A phase 1 study of anti-TGFbeta receptor type-II monoclonal antibody LY3022859 in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2017 Apr;79(4):673-680. doi: 10.1007/s00280-017-3245-5. Epub 2017 Mar 9. PMID 28280971

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants that completed Cohort 1A, Cohort 1B or Cohort 2 are those who died, had progressive disease (PD) or off treatment & censored due to study completion.
Groups:
- 1.25 mg/kg LY3022859: Cohort 1A: 1.25 milligram/kilogram (mg/kg) LY3022859 administered intravenously (IV) once every 2 weeks (Q2W) during 6-week treatment cycles.
- 12.5 mg LY3022859: Cohort 1B: 12.5 mg IV once Q2W during 6-week treatment cycles.
- 25 mg LY3022859: Cohort 2: 25 mg IV once Q2W during 6-week treatment cycles.
Period: Overall Study
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859
Started | 2 | 5 | 7
Received at Least One Dose of Study Drug | 2 | 5 | 7
Completed | 0 | 3 | 6
Not Completed | 2 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician's Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859 | Total
Number analyzed (Participants) | 2 | 5 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (19.09) | 62.2 (9.44) | 55.0 (16.80) | 59.1 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 2 | 3 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 0 | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 5 | 7 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 5 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as an AE occurring during Cycle 1(first 6 weeks of treatment) that was considered at least possibly related to study drug, was considered dose-dependent, and fulfilled a criteria selected (using the National Cancer Institute Common Terminology Criteria for Adverse Events,version 4.0 [NCI-CTCAE v 4.0] [NCI 2009]):Grade(Gr)≥3 nonhematological toxicity,Gr4 thrombocytopenia lasting at least 5 days and/or complicated with bleeding,Gr≥3 febrile neutropenia(ntr),Gr4 ntr of >5 days' duration,increase(incr)of at least 1 gr from a preexisting Gr1 valvular insufficiency or any new Gr≥2 valvular toxicity,left ventricular(vtr) ejection fraction decrease of 10% in absolute value or 16% in relative value,incr in right vtr systolic pressure dysfunction from mild to moderate(mod) or from mod to severe,incr in left atrial or ventricular chamber size of ≥2 cm and ≥1cm respectively,any other life-threatening toxicity,significant morphologic on cardiac echocardiogram,any major ocular.
Time Frame: First Dose Up to 6 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 2 | 5 | 7
Participants | 2 | 0 | 2

2. Secondary Outcome: Maximum Tolerated Dose (MTD) of IMC-TR1
Description: The MTD was defined as the highest dose level at which ≤33% of participants experienced a DLT during Cycle 1.
Time Frame: First Dose through Cycle 1 (6 Weeks)
Population: All participants who received at least one dose of study drug and completed cycle 1 or discontinued treatment due to a DLT during the cycle 1.
Measure: Number; unit: milligram (mg)
Groups:
- All Participants Receiving a Flat Dose: 12.5 mg LY3022859 Cohort 1B: 12.5 mg IV once Q2W during 6-week treatment cycles.
  25 mg LY3022859 Cohort 2: 25 mg IV once Q2W during 6-week treatment cycles.
Arm/Group | All Participants Receiving a Flat Dose
Number analyzed (Participants) | 3
milligram (mg) | NA — MTD was not reached.

3. Secondary Outcome: Maximum Tolerated Dose (MTD) of IMC-TR1 (1.25 mg/kg LY3022859 ) for Participants Receiving a Weight-Based Dose
Description: The MTD was defined as the highest dose level at which ≤33% of participants experienced a DLT during Cycle 1.
Time Frame: First Dose through Cycle 1 (6 Weeks)
Population: as for outcome 2
Measure: Number; unit: milligram/kilogram (mg/kg)
Groups:
- All Participants Receiving a Weight-Based Dose: 1.25 mg/kg LY3022859 Cohort 1A: 1.25 milligram/kilogram (mg/kg) LY3022859 administered intravenously (IV) once every 2 weeks (Q2W) during 6-week treatment cycles.
Arm/Group | All Participants Receiving a Weight-Based Dose
Number analyzed (Participants) | 2
milligram/kilogram (mg/kg) | NA — MTD was not reached.

4. Secondary Outcome: Number of Dose-Limiting Toxicities (DLTs)
Time Frame: First Dose through Cycle 1 (6 Weeks)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: DLTs
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 2 | 5 | 7
DLTs | 2 | 0 | 2

5. Secondary Outcome: Immunogenicity - Development of Antibodies Against IMC-TR1
Time Frame: Cycle 1 - Day 1 and Day 29, Cycle 2 - Day 15, Cycle 3 and Each Consecutive Cycle - Day 1
Population: Zero participants were analyzed. Immunogenicity data were not collected.
Groups:
- 25 mg LY3022859: Cohort 2: 25mg IV once Q2W during 6-week treatment cycles.
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR]) (Antitumor Activity of IMC-TR1 as Monotherapy, Assessed Via Tumor Measurement by Response Evaluation Criteria in Solid Tumors, Version 1.1)
Description: ORR is the best response of CR or PR as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: First Dose to Measured Progressive Disease (Up To 21.3 Weeks)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 2 | 5 | 7
percentage of participants | 0 [0 to 84.2] | 0 [0 to 52.2] | 0 [0 to 41.0]

7. Secondary Outcome: Pharmacokinetics (PK) - Area Under the Concentration-time Curve (AUC[0-tlast]) and AUCτ of IMC-TR1
Description: AUC (0-tlast) is area under the concentration versus time curve from the time zero to tlast.
  AUCτ is area under the concentration versus time curve during 1 dose interval (336 hours).
Time Frame: Cycle (C) 1 Day (D) 1: 1, 2, 4, 8 hours (h); C1 D2: 24 h; C1 D3: 48 h; C1 D5: 96 h; C1 D8: 168 h; C1 D15: 336 h; C2 D15: 1, 2, 4, 8 h; C2 D16: 24 h; C2 D17: 48 h; C2 D19: 96 h; C2 D22: 168 h, C2 D29: 336 h
Population: All participants who received at least one dose of study drug and had evaluable PK data. PK of LY3022859 was not characterized at the 1.25-mg/kg dose level because of infusion interruptions thus no data collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(µg·hr/mL)
Arm/Group | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 5 | 5
microgram*hour per milliliter(µg·hr/mL)
  Cycle 1 (AUC[0-tlast]) | 28.5 (18) | 60.2 (30)
  Cycle 2 (AUCτ): number analyzed (Participants) | 0 | 3
  Cycle 2 (AUCτ) |  | 60.7 (35)

8. Secondary Outcome: Pharmacokinetics - Maximum Concentration (Cmax) of IMC-TR1
Time Frame: as for outcome 7
Population: All participants who received at least one dose of study drug and had evaluable PK data. PK of LY3022859 was not characterized at the 1.25 mg/kg dose level because of infusion interruptions thus no data collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 5 | 5
microgram per milliliter (µg/mL)
  Cycle 1 | 4.34 (9) | 5.10 (21)
  Cycle 2: number analyzed (Participants) | 2 | 3
  Cycle 2 | 3.52 (9) | 5.01 (28)

9. Secondary Outcome: Pharmacokinetics - Minimum Concentration (Cmin) of IMC-TR1
Description: Pharmacokinetics - Minimum concentration (Cmin) of IMC-TR1
Time Frame: Cycle 2 Day 1: Prior to fourth infusion 0 hour (h)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | 12.5 mg LY3022859 | 25 mg LY3022859
Number analyzed (Participants) | 2 | 3
microgram/milliliter (µg/mL) | NA (NA) — Concentrations were below the limit of quantification. | NA (NA) — Concentrations were below the limit of quantification.

ADVERSE EVENTS:
Groups:
- 12.5 mg LY3022859: Cohorts 1B: 12.5 mg IV once Q2W during 6-week treatment cycles.
- 25 mg LY3022859: Cohorts 2: 25 mg IV once Q2W during 6-week treatment cycles.
Arm/Group | 1.25 mg/kg LY3022859 | 12.5 mg LY3022859 | 25 mg LY3022859
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/5 | 4/7
Other Adverse Events (participants affected / at risk) | 2/2 | 4/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.25 mg/kg LY3022859 (N=2) | 12.5 mg LY3022859 (N=5) | 25 mg LY3022859 (N=7)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.25 mg/kg LY3022859 (N=2) | 12.5 mg LY3022859 (N=5) | 25 mg LY3022859 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 3 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Maximum Tolerated Dose (MTD) was not reached. Dose escalation beyond 25 mg LY3022859 was not completed due to DLT. Two participants who received 1.25 mg/kg required permanent interruption of administration because they developed DLT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days